CLINICAL TRIAL: NCT03812354
Title: THRIVE (Transnasal Humidified Rapid Insufflation Ventilatory Exchange) in Children at Different Flow Rates
Brief Title: THRIVE in Children at Different Flow Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Thomas Riva, Consultant Anaesthesia, MD, Principal investigator, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Riva2018
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Apnea; Ventilation Therapy; Complications
Keywords: infant; airway management; apneic oxygenation
MeSH Terms: conditions — Apnea | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE 2L/kg/min using OptiFlow (Active Comparator): High-flow nasal cannula therapy with 2L/kg/min with 100% oxygen via OptiFlow by Fisher&Paykel, Auckland, New Zealand.
  Interventions: Other: THRIVE 2L/kg/min
- THRIVE 4L/kg/min using OptiFlow (Experimental): After apnea sets in and mask ventilation is successfully established, randomization envelopes are opened and according to group allocation, the following oxygen delivery system is applied.
  High-flow nasal cannula therapy with 4L/kg/min with 100% oxygen via OptiFlow by Fisher&Paykel, Auckland, New Zealand.
  Interventions: Other: THRIVE 4L/kg/min

INTERVENTIONS:
Other: THRIVE 4L/kg/min — High-flow nasal cannula therapy with 4L/kg/min with 100% oxygen via OptiFlow by Fisher&Paykel, Auckland, New Zealand.
  Other Names: Optiflow
  Arms: THRIVE 4L/kg/min using OptiFlow
Other: THRIVE 2L/kg/min — High-flow nasal cannula therapy with 2L/kg/min with 100% oxygen via OptiFlow by Fisher&Paykel, Auckland, New Zealand.
  Other Names: Optifloe
  Arms: THRIVE 2L/kg/min using OptiFlow

SUMMARY:
This study investigates under controlled circumstances the concept of THRIVE to improve the ventilation and the carbon dioxide elimination, to prolong the apnoea time without deoxygenation and to improve safety of airway management in pediatric patients.

DETAILED DESCRIPTION:
Eligible, consented children will be prepared for general anaesthesia in the usual way. After start of anesthesia (="induction"), adequate face-mask ventilation will be established. The sealed envelope for randomisation will then be opened. Standard anesthesia will be continued, either using sevoflurane or propofol (anesthesia depth controlled by Narcotrend, to measure anesthesia depth using processed EEG waves). They will receive additional non-invasive monitoring for this study, such as transcutaneous measurement of tcCO2 and O2, NIRS, and thoracic electrical impedance tomography (EIT, PulmoVista® 500, Draeger, Luebeck, Germany) All patients will receive neuromuscular blockade medication of 2 x ED95 (standard intubation dose) to facilitate airway management and total intravenous anesthesia will be installed (continuous application of i.v. anesthesia medication). Up to two minutes of bag-mask ventilation with 100% oxygen and flow rates of 6-8L/min will be applied until an expired oxygen concentration of >90% is reached, as well as an SpO2 of 100% and an transcutaneous CO2 of 30-40mmHg.

For the study intervention, the bag-mask ventilation will be discontinued, and the child will be left apnoeic (the same happens always during intubation) until the saturation drops to 95%, which is still a low normal value. According randomization, any of the two study intervention s will be applied (THRIVE therapy with 100% O2 2l/kg/min, THRIVE therapy with 100% O2 4l/kg/min, all via nasal cannulas) while simultaneously guaranteeing an open airway by using Esmarch's procedure (jaw thrust) and an oral airway (Guedel tube). ECG, pulse-oximetry, blood pressure, Narcotrend, NIRS, thoracic EIT, PtcO2, PtcCO2 will be measured continuously over the study period. The time until desaturation from SpO2 100% to SpO2 95% will be also measured. A chest ultrasound at the end of the intervention will prove that no pneumothorax developed during the procedure. The study intervention will end at the time the saturation reaches SpO2 95% or when any other break-up criteria are reached. Bag mask ventilation will then be re-applied until SpO2 reaches again 100% and the patient will be treated according to the attending anaesthesiologist to ultimately establish a patent airway. Break-up criteria during apnoea are: SpO2 below 95%, transcutaneous CO2 above 70 mmHg, or time of apnoea >10 minutes. Drop of NIRS > 30% from baseline. A postmedication interview will be performed before PACU discharge.

ELIGIBILITY:
Inclusion Criteria:

* paediatric patients undergoing elective surgery requiring general anesthesia with intubation at the University Hospital - Inselspital in Bern.
* ASA physical status 1&2
* 10-15kg
* legal guardians providing written informed consent.

Exclusion Criteria:

* known or suspected difficult intubation
* oxygen dependency
* congenital heart or lung disease
* obesity BMI>20kg/m2
* high aspiration risk (requiring rapid sequence induction intubation).

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change of tcCO2 in mmHg/min | 10 minutes
  mean tcCO2 increase in mmHg/min during apnoea time, measured transcutaneously.

SECONDARY OUTCOMES:
desaturation from SpO2 100% to 95% | 10 minutes
  time (in seconds) until desaturation from SpO2 100% to 95%
tcO2 in mmHg/min | 10 minutes
  Changes in tcO2 in mmHg/min
NIRS | 10 minutes
  changes in brain oxygenation (measured by near infrared spectroscopy (NIRS)) during apnoea time
Electrical impedance tomography | 10 minutes
  changes in electrical impedance tomography (EIT) to validate ventilatory effect

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD, Study Chair — Department of Anesthesia, University Hospital Bern
Locations (2):
- Switzerland (2):
  - Inselspital, Bern
  - University Hospital Bern, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riva T, Preel N, Theiler L, Greif R, Butikofer L, Ulmer F, Seiler S, Nabecker S. Evaluating the ventilatory effect of transnasal humidified rapid insufflation ventilatory exchange in apnoeic small children with two different oxygen flow rates: a randomised controlled trial. Anaesthesia. 2021 Jul;76(7):924-932. doi: 10.1111/anae.15335. Epub 2020 Dec 22. PMID 33351194